CLINICAL TRIAL: NCT03544463
Title: A Prospective, Self-controlled, First-night Order Cross-over and Evaluator-blind Pivotal Study to Evaluate the Efficacy and Safety of the iNAP® Sleep Therapy System in Adults With Obstructive Sleep Apnea (OSA)
Brief Title: Pivotal Study of the iNAP® in Adults With OSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Somnics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: iNAP®-TW-1701
Record Dates: First submitted 2018-03-15; First posted 2018-06-01 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treated (Experimental): iNAP® Sleep Therapy System Treatment Intervention
  Interventions: Device: iNAP® Sleep Therapy System
- Baseline/Control (No Intervention): Self-controlled, pre-treatment baseline condition

INTERVENTIONS:
Device: iNAP® Sleep Therapy System — The iNAP® provides a pressure gradient within the oral cavity, which pulls the tongue toward the upper palate and pulls the soft palate forward in a way that enhances the patency of the upper airway near the pharynx so that upper airway patency can be maintained to prevent sleep-disordered breathing.
  Arms: Treated

SUMMARY:
A Prospective, Self-controlled, First-night Order Cross-over and Evaluator-blind Pivotal Study to Evaluate the Efficacy and Safety of iNAP® Sleep Therapy System in Adults with Obstructive Sleep Apnea (OSA)

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) impacts sleep quality of patients, which contributes significantly to hypertension, stroke, myocardial infarction and other health problems. Intraoral devices, such as tongue retaining devices, palatal lifting devices and mandibular repositioning devices designed to increase the patency of the airway and to decrease airway obstruction, are used to treat OSA. To this end, the investigators are conducting a prospective, self-controlled, first-night order cross-over and evaluator-blind pivotal study to evaluate the efficacy and safety of iNAP® Sleep Therapy System (iNAP®), a tongue and soft palate retaining intraoral device, in adults with OSA.

ELIGIBILITY:
Inclusion Criteria:

* Patients able to read and sign on the informed consent form and able to comply with study requirements.
* Body mass index (BMI) <33 kg/m2
* AHI between 15~55
* Pass a device feasibility test

Exclusion Criteria:

* Obstructed nasal passages
* Hypoxemia (SpO2 <80%)
* Primary insomnia or other suspected sleep disorder other than OSA
* Muscle diseases, e.g. CSA
* Patients with potential complications of sleep apnea that, in the opinion of the Investigator, may affect the study interpretation or the health or safety of the patients

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-06-06 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
iNAP®-treated response rate over the apnea-hypopnea index (AHI)* | first treatment night
  *AHI is the number of apnea/hypopnea events divided by total sleep time (TST), i.e., the number of hours of sleep. The reduction rate of AHI is calculated by dividing the AHI reduction on the Tx PSG Study when compared to the Baseline PSG Study with individual baseline AHI. An AHI reduction rate of 50% is considered responsive, namely, responder. Therefore, an overall ratio of responder to the primary endpoint cohort is the response rate.

SECONDARY OUTCOMES:
Clinical Global Impression of Change (CGI-C) | first treatment night
  Global impression changes as rated by the physicians
Negative pressure maintenance time (hr) | first treatment night
  The time period of iNAP® in providing effective negative pressure within the oral cavity
Change of Oxygen Desaturation Index (ODI)** from the Baseline PSG Study compared to the Tx PSG Study | first treatment night
  **ODI is the event number of oxygen level drops by 3 percent or more from baseline divided by total sleep time (TST), i.e., the number of hours of sleep.

OTHER OUTCOMES:
Number of participants with abnormal laboratory values and/or adverse events in this entire study. | through study completion, up to 8 weeks
  All safety events will be listed and tabulated for their occurrence rate

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Mo Lin, Principal Investigator — Shin Kong Wu Ho-Su Memorial Hospital
Locations (1):
- Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No